CLINICAL TRIAL: NCT03796039
Title: Stand if You Can- A Randomized Control Trial
Brief Title: Stand if You Can: A Standing Intervention in Long Term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Horizon Health Network (Other); St. Thomas University (Other); Universite de Moncton (Other); Canadian Frailty Network (Other)
Responsible Party: Principal Investigator, Danielle Bouchard, Associate Investigator, University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CAT2018-15
Record Dates: First submitted 2018-12-20; First posted 2019-01-08 (Actual); Results first posted 2021-07-06 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Frailty; Sedentary Behavior; Physical Disability
Keywords: Long Term Care; Physical Function
MeSH Terms: conditions — Frailty; Sedentary Behavior | interventions — Standing Position

STUDY DESIGN:
Intervention Model Description: Long term care (LTC) facilities will be recruited, with half of the LTC facilities randomized as the intervention (n=2) and half as the control group (n=2).
Who Masked: Investigator
Masking Description: Investigator was masked at pre-testing. It was unknown which participants would be receiving the intervention. However, due to resources this was not repeated at post testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standing and Social Intervention (Experimental): Participants be exposed to an additional 100 minutes of standing per week. Participants will do this by standing for 20 minutes Monday through Friday.
  Interventions: Behavioral: Standing
- Control Group (No Intervention): Control group will receive social visits, but no exposure to standing

INTERVENTIONS:
Behavioral: Standing — Standing for an additional 100 minutes per week; 20 minutes Monday-Friday
  Arms: Standing and Social Intervention

SUMMARY:
It is currently unknown if reducing sitting time, an activity that is highly prevalent in frail older adults living in long term care (LTC) facilities, is associated with an improvement in physical capacity such as walking speed. Simple tasks such as walking speed is associated with important outcomes for residents in LTC such as autonomy and hospitalization. The investigators hypothesize that standing an additional 100 minutes per week for 5 months will result in a clinically meaningful improvement in walking speed (0.1m/sec) in LTC residents compared to residents receiving a sitting social activity.

DETAILED DESCRIPTION:
LTC facilities from Moncton and Fredericton will be recruited, with half of the LTC facilities randomized as the intervention and half as the control group. The investigators are aiming to enrol half of the LTC in Fredericton and half in Moncton. A total of 88 residents (44 in the control group, 44 in the intervention group) will be enrolled in the program.

ELIGIBILITY:
Inclusion Criteria:

* Resident at one of the selected LTC facilities;
* Able to provide consent or have a power of attorney agree on behalf of a resident to participate in the study;
* Able to walk for ten meters, with or without a walking aid; The main outcome is walking speed performed for a distance of 10 meters. Therefore, we want everyone who participates in the study to be able to complete the test at baseline. This way we can answer the main research question, while adhering to our sample size calculation.

Exclusion Criteria:

* If Identified by staff at the facility as too high risk for falling by participating in the intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pine Grove Nursing Home, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooling K, Bouchard DR, Gallibois M, Hebert J, Senechal M, Jarrett P, McGibbon C, Richard E, Handrigan G. Stand if you can- A parallel, superiority cluster randomized controlled trial to improve gait speed for long term care residents. JAR Life. 2025 May 9;14:100015. doi: 10.1016/j.jarlif.2025.100015. eCollection 2025. PMID 40469490

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standing and Social Intervention | Control Group
Started | 50 | 47
Completed | 41 | 42
Not Completed | 9 | 5
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standing and Social Intervention | Control Group | Total
Number analyzed (Participants) | 50 | 47 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 87.14 (8.46) | 85.11 (7.63) | 86 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 68
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.93 (6.53) | 25.56 (9.01) | 26.2 (7.8)
Frailty [Mean (Standard Deviation); unit: units on a scale] — Frailty was measured using the Clinical Frailty Scale (1-9). 1 indicates very fit, 9 indicates terminally ill. LTC staff were asked to rate participants at pre and post intervention
  units on a scale | 6 (1.5) | 6.13 (0.8) | 6.1 (1.2)
Transfer Status (Independent Transfer) [Count of Participants; unit: Participants] — Transfer status was assessed by LTC staff following jurisdiction regulations (Work Safe New Brunswick). It is assessed upon admission, quarterly (90 days) and when a significant change in health status occurs (e.g., fall, stroke). For our study, we used the most recent Transfer status update. Residents were categorized as requiring no assistance to transfer from sit to stand (independent), requiring staff assistance to stand (assisted transfer), or requiring staff and mechanical assistance to stand (dependent).
  Participants | 8 | 25 | 33
Length of stay in LTC [Mean (Standard Deviation); unit: years] | 4.6 (5.4) | 3.9 (3.5) | 4.2 (4.5)
Cognition (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The mini-mental state examination was administered by research assistants at baseline to assess cognition. Scored out of 30, the questionnaire categorized a person as having none, mild or severe cognitive impairment. A score of 0-17 indicates severe cognitive impairment, 18-23 as mild, and 24-30 as no cognitive impairment.
  units on a scale | 15.76 (9.2) | 17.7 (8.8) | 16.7 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Walking Speed
Description: Measured by the 10m walking speed test
Time Frame: Pre and post intervention testing
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 50 | 47
m/s
  Pre | 0.34 (0.17) | 0.43 (0.20)
  Post | 0.35 (0.20) | 0.40 (0.20)

2. Secondary Outcome: Change in Balance
Description: Measured by a portable device (Wii Balance board), which has sensors that detects sway .
Time Frame: Pre and post testing (following the 5 month intervention). Data was collected but investigators are still analyzing findings.
Reporting Status: Not Posted, anticipated posting 2024-09

3. Secondary Outcome: Change in Leg Strength
Description: Using hand-held dynamometer to quantify leg strength through knee extension
Time Frame: Pre-Post Testing (following the 5 month intervention)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 50 | 47
kg
  Pre | 9.48 (5.95) | 7.87 (5.42)
  Post | 9.15 (5.25) | 7.28 (4.90)

4. Secondary Outcome: Change Lower Limb Power
Description: Using the 30second sit-stand test following senior fitness test protocol
Time Frame: Pre-Post Testing (following the 5 month intervention)
Measure: Mean (Standard Deviation); unit: Number of repetitions
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 50 | 47
Number of repetitions
  Pre | 0.74 (1.84) | 0.89 (2.34)
  Post | 0.71 (1.81) | 1.1 (2.82)

5. Secondary Outcome: Change in Anxiety Symptoms
Description: The Geriatric Anxiety Inventory (Scale 0-20). A low score means a better outcome.
Time Frame: Pre-Post Testing (following the 5 month intervention)
Population: Only participants with MMSE score greater than or equal to 18 were included (to ensure participants had the cognitive abilities to respond to the questionnaires)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 20 | 25
units on a scale
  Pre | 6.1 (7.2) | 6.6 (6.0)
  Post | 6.7 (7.1) | 6.6 (6.1)

6. Secondary Outcome: Depression
Description: Geriatric Depression Scale Short Form (0-15 scale). Lower score is better outcome.
Time Frame: Pre-Post Testing (following the 5 month intervention)
Population: Only participants with a MMSE score of 18 or higher were included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 20 | 25
score on a scale
  Pre | 5.1 (3.2) | 4.9 (3.5)
  Post | 5.5 (4.0) | 4.5 (2.9)

7. Secondary Outcome: Loneliness
Description: Loneliness was measured using the UCLA Loneliness Scale (20-80). A low score indicates a better outcome
Time Frame: Pre-Post Testing (following the 5 month intervention)
Population: Participants only included if MMSE score is equal to or greater than 18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 20 | 25
score on a scale
  Pre | 42.3 (12.0) | 39.7 (12.6)
  Post | 38.7 (12.4) | 33.8 (11.2)

8. Secondary Outcome: Fall Efficacy
Description: Falls Efficacy Scale-International Questionnaire (16-64 scale). Low score indicates a better score
Time Frame: Pre-Post Testing (following the 5 month intervention)
Population: This was only measured among participants who had a MMSE score of 18 or higher (to ensure they had the cognitive capacity to properly answer the questionnaire)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 20 | 25
score on a scale
  Pre | 36.7 (13.2) | 31.0 (12.8)
  Post | 41.3 (17.4) | 39.0 (11.8)

9. Secondary Outcome: Rate of Falls
Description: Falls, injuries due to falls and hospitalization will be collected at 3 timepoints
Time Frame: The number of falls will be collected from three timeframes: 1. Between 6 months prior to and the start of program 2. the duration of the program (5 months) 3. From the end of the program to 6 months follow up. Data is still being analyzed at this time.
Reporting Status: Not Posted, anticipated posting 2024-09

10. Secondary Outcome: Metabolic Profile - Triglycerides
Description: Capillary blood analyzed with a cardiochek device. Blood collected via a finger prick and analyzed with a cardiochek device. Note that Total Cholesterol, HDL, Triglycerides, LDL and Glucose were all measured using the cardiochek device.
Time Frame: Pre-Post Testing (before and following the 5 month intervention).
Population: Blood draws were difficult among this population due to participant agitation, therefore we were not able to collect blood for all participants
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 32 | 38
mmol/L
  Pre | 1.79 (1.30) | 1.21 (0.45)
  Post | 1.48 (0.74) | 1.47 (0.82)

11. Secondary Outcome: Social Behaviours
Description: Semi-structured interviews with residents (participants and non-participants), family members and staff will be administered at the end of the study
Time Frame: Pre-Post Testing (following the 5-month intervention). Data has been collected, but is still being analyzed
Reporting Status: Not Posted, anticipated posting 2024-09

12. Secondary Outcome: Metabolic Profile - High Density Lipoprotein Cholesterol
Description: High Density Lipoprotein (HDL) cholesterol was analyzed using the CardioChek Professional Analyzer system (PTS Diagnostics, Whitestown, Indiana, USA). A finger prick was conducted using a single use lancet and approximately 60 µL of whole blood was collected for this test.
Time Frame: Pre and post testing (before and after the 5-month intervention)
Population: Research assistants were not able to collect blood data for all participants (due to participant agitation or refusal)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 32 | 38
mmol/L
  Pre | 1.37 (1.52) | 1.33 (0.51)
  Post | 1.27 (0.44) | 1.17 (0.57)

13. Secondary Outcome: Metabolic Profile - Low Density Lipoprotein Cholesterol
Description: Low-density lipoprotein was assessed using a CardioChek Professional Analyzer system (PTS Diagnostics, Whitestown, Indiana, USA).
Time Frame: Pre-Post intervention (before and after 5-month intervention)
Population: Research assistants were not able to collect blood data for all participants (due to participant agitation or refusal)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 32 | 38
mmol/L
  Pre | 2.40 (1.63) | 2.91 (1.42)
  Post | 2.19 (1.21) | 2.72 (1.56)

14. Secondary Outcome: Metabolic Profile - Blood Glucose
Description: Fasted blood glucose was analyzed using a CardioChek Professional Analyzer system (PTS Diagnostics, Whitestown, Indiana, USA).
Time Frame: Pre-Post Intervention (before and after 5-month intervention)
Population: Research assistants were not able to collect blood data for all participants (due to participant agitation or refusal)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standing and Social Intervention | Control Group
Number analyzed (Participants) | 32 | 38
mmol/L
  Pre | 5.96 (2.38) | 5.43 (1.95)
  Post | 6.08 (2.29) | 5.47 (1.77)

ADVERSE EVENTS:
Time Frame: During trial (5 months)
Arm/Group | Standing and Social Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/47
Other Adverse Events (participants affected / at risk) | 1/50 | 0/47
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standing and Social Intervention (N=50) | Control Group (N=47)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03796039/Prot_SAP_000.pdf